CLINICAL TRIAL: NCT03881995
Title: Effect of Insulin Glargine and Lixisenatide Versus Insulin Glargine on Brain Insulin Sensitivity in Patients With Type 2 Diabetes
Brief Title: Effects of Insulin Glargine and Lixisenatide on the Brain
Acronym: Lixibrain01
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 808/2018AMG1; 2018-003557-21 (EudraCT Number)
Record Dates: First submitted 2019-02-19; First posted 2019-03-20 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iGlarLixi (Active Comparator): Subjects will receive premixed Insulin glargine + lixisenatide once daily for 12 weeks
  Interventions: Drug: IGlarLixi
- Insulin glargine (Active Comparator): Subjects will receive Insulin glargine once daily for 12 weeks
  Interventions: Drug: Insulin Glargine 100 UNT/ML

INTERVENTIONS:
Drug: IGlarLixi — Dose titration will be done based on the subjects fasting blood glucose
  Arms: iGlarLixi
Drug: Insulin Glargine 100 UNT/ML — Dose titration will be done based on the subjects fasting blood glucose
  Arms: Insulin glargine

SUMMARY:
1. Background During the last years, the brain has been identified as a major insulin-sensitive organ . The investigators and also other scientists identified hypothalamus, fusiform gyrus and prefrontal cortex as major insulin-sensitivity brain areas in humans . Brain insulin action regulates important physiological functions in humans such as food intake, body weight regulation, and cognition. Furthermore, animal studies suggest that insulin action specifically in the brain is involved in the control of peripheral glucose metabolism via regulation of the sensitivity to insulin in the rest of the body. Recently, the investigators were able to replicate these findings in humans: The investigators measured whole-body insulin sensitivity in combination with the well-established experimental delivery of human insulin to the brain via an intranasal approach. Peripheral insulin sensitivity was profoundly improved by brain insulin action in lean but not in obese healthy volunteers. What determines the effectiveness of this brain-derived pathway is still unknown. Furthermore, insulin resistance of the brain is linked to neurodegenerative diseases possibly explaining the elevated risk for such diseases in patients with type 2 diabetes.

   GLP-1 receptor agonists have been shown to acutely modulate appetite- and reward-related brain areas in humans. Research in animals suggest a close interaction between insulin and GLP-1 action especially in homeostatic centers of the hypothalamus. In this context, it is important that GLP-1 sensitivity of the brain is still present in the insulin resistant human brain.

   The investigators therefore hypothesized that GLP-1 agonists are able to improve insulin sensitivity of the brain; this might be one mechanism how GLP-1 agonists lead to weight loss and improved glucose metabolism. This might also have beneficial implications for cognitive function.

   However, at present, there are no human studies examining the effect of a GLP-1 agonist on brain activity and especially insulin action in the brain in patients with type 2 diabetes mellitus (T2D).

   Furthermore, there is no study in humans examining the effect of newly initiated insulin therapy on brain activity and especially insulin action in the brain in patients with T2D.
2. Rationale Based on the close interplay between hypothalamic insulin and GLP-1 signalling, the investigators hypothesize that the antidiabetic therapy with insulin glargine/lixisenatide combination (iGlarLixi) induces improved hypothalamic and prefrontal insulin sensitivity compared to a therapy with insulin glargine alone. This could underlay iGlarLixi's beneficial effects on body weight and whole-body glucose homeostasis.
3. Objective To assess whether treatment with iGlarLixi versus insulin glargine changes brain regional insulin sensitivity and thereby glucose metabolism, eating behaviour, and cognition in patients with type 2 diabetes insufficiently controlled with oral antidiabetic drugs (OAD).

ELIGIBILITY:
Inclusion Criteria:

* Must be between 18 and 65 years at the time of signing the informed consent.
* BMI 25-45 kg/m²
* Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures.
* Ability to adhere to the study visit schedule and other protocol requirements.
* Patients with type 2 diabetes mellitus diagnosed for at least 1 year before the screening visit (visit 1) treated for at least 3 months prior to visit 1 with only metformin or metformin and a sodium glucose co-transporter 2 inhibitor, and patients who are not adequately controlled with this treatment.
* Females of childbearing potential (FCBP) must agree

  * to utilize a highly effective forms of contraception (Pearl index < 1) or practice complete abstinence from heterosexual contact while participating in the study (including dose interruptions), and for at least 28 days after study treatment discontinuation and must agree to pregnancy testing during this timeframe
  * to abstain from breastfeeding during study participation and 28 days after study drug discontinuation.
* Males must agree

  * to use a latex condom during any sexual contact with FCBP while participating in the study and for 28 days following discontinuation from this study, even if he has undergone a successful vasectomy
  * to refrain from donating semen or sperm while participating in this study and for 28 days after discontinuation from this study treatment.
* All subjects must agree to refrain from donating blood while on study drug and for 28 days after discontinuation from this study treatment.
* All subjects must agree not to share medication.

Exclusion Criteria:

* HbA1c at screening visit less than 7.5% or more than 12% for patients previously treated with metformin alone or with metformin and a second oral anti-diabetic treatment.
* Women during pregnancy and lactation.
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal products. This includes iGlarLixi, insulin glargine, and human nasal insulin.
* Use of oral glucose-lowering agents other than those stated in the inclusion criteria or any injectable glucose-lowering agents during 3 months before screening
* History of discontinuation of a previous treatment with a GLP-1 receptor agonist (GLP-1 RA) due to safety/tolerability issue or lack of efficacy.
* Patient who has previously participated in any clinical trial with lixisenatide or the insulin glargine + lixisenatide fixed ratio combination or has previously received lixisenatide.
* Any contraindication to metformin use, according to local labeling.
* Use of weight loss drugs within 3 months prior to screening visit.
* Within the last 6 months prior to screening visit: myocardial infarction, unstable angina, or heart failure requiring hospitalization. Planned coronary, carotid or peripheral artery revascularisation procedures to be performed during the study period.
* History of stroke.
* History of pancreatitis (unless pancreatitis was related to gallstones and cholecystectomy was already performed), chronic pancreatitis, pancreatitis during a previous treatment with incretin therapies, pancreatectomy, stomach/gastric surgery.
* Personal or immediate family history of medullary thyroid cancer (MTC) or genetic conditions that predispose to MTC (eg, multiple endocrine neoplasia syndromes).
* Uncontrolled or inadequately controlled hypertension (systolic blood pressure above 160 mmHg or diastolic blood pressure above 90 mmHg) at screening visit.
* At screening visit, Body Mass Index (BMI) less than or equal to 25 or above 45 kg/m².
* At screening visit ALT or AST more than 3 ULN.
* At screening visit calcitonin above or equal to 20 pg/mL (5.9 pmol/L).
* Exclusion Criteria for randomization at the end of the screening period:

  * HbA1c less than 7.5% or above 12%.
  * Amylase and/or lipase more than 3 ULN.
  * Calcitonin above or equal to 20 pg/mL (5.9 pmol/L).
* Participation in other clinical trials or observation period of competing trials up to 30 days prior to this study.
* Known malformation of the central nervous system
* Persons working nightshift
* Treatment with drugs with central nervous actions or systemic steroid therapy
* Any relevant (according to investigator's judgment) cardiovascular disease, e.g. myocardial infarction, acute coronary syndrome, unstable angina pectoris, PTCA, heart failure (NYHA II-IV), planned coronary, carotid or peripheral artery revascularisation procedures to be performed during the study period.
* Indication of liver disease, as per medical history or defined by serum levels of either Alanine Aminotransferase (ALT [SGPT]), Aspartate Aminotransferase (AST [SGOT]), or Alkaline Phosphatase above 3 x upper limit of normal (ULN) as determined during screening.
* Alcohol abuse, defined as more than 20 gr/day
* Impaired renal function, defined as estimated Glomerular Filtration Rate (eGFR) ≤ 60 ml/min (MDRD formula) as determined during screening.
* Known structural and functional urogenital abnormalities that that predispose for urogenital infections.
* Subjects with a haemoglobin (Hb) between 14 and 18 g/dl (for males) and Hb between 12 and 16 g/dl (for females) at screening.
* Bariatric surgery within the past two years and other gastrointestinal surgeries that induce chronic malabsorption within the last 5 years.
* Medical history of cancer (except for basal cell carcinoma) and/or treatment for cancer within the last 5 years.
* Treatment with anti-obesity drugs 3 months prior to informed consent or any other treatment at the time of screening (i.e. surgery, aggressive diet regimen, etc.) leading to unstable body weight.
* Known autoimmune disease (except autoimmune disease of the thyroid gland) or chronic inflammatory condition.
* Claustrophobia
* Any other clinically significant major organ system disease at screening such as relevant gastrointestinal, neurologic, psychiatric, endocrine (i.e. pancreatic), hematologic, malignant, infection or other major systemic diseases making implementation of the protocol or interpretation of the study results difficult.
* Presence of any contraindication for the conduct of an MRI investigation, such as cardiac pacemakers, ferromagnetic haemostatic clips in the central nervous system, metallic splinters in the eye, ferromagnetic or electronically operated active devices like automatic cardioverter defibrillators, cochlear implants, insulin pumps and nerve stimulators, prosthetic heart valves etc.
* Any other clinical condition that would jeopardize subjects' safety while participating in this clinical trial.
* Refusal to get informed of unexpected detected pathological MRI findings
* History of diabetic ketoacidosis
* Severe gastric or bowel disease (including gastroparesis)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-29 (Actual)

PRIMARY OUTCOMES:
Brain insulin sensitivity | Change from baseline brain insulin sensitivity at 12 weeks
  Effect of 12 weeks treatment with iGlarLixi or Glargine on brain insulin sensitivity assessed by functional magnetic resonance imaging (fMRI) as change in regional cerebral blood flow (rCBF) from before to 30 minutes after nasal insulin spray application.

SECONDARY OUTCOMES:
Processing of food pictures | Change from baseline processing of food pictures at 12 weeks
  Effect of 12 weeks treatment with iGlarLixi or Glargine on resting state brain activity and on brain response to food pictures and control pictures as assessed by functional magnetic resonance imaging.
Cognitive function | Change from baseline participant's speed of response and the accuracy of pointing at 12 weeks
  Effect of 12 weeks treatment with iGlarLixi or Glargine on cognitive function assessed by established Motor Screening Task (MOT). Outcome measures: assess the participant's speed of response and the accuracy of pointing.
  It is part of Cambridge Neuropsychological Test Automated Battery (CANTAB) to assess neurocognition. All CANTAB tests are evaluated together.
Cognitive function | Change from baseline reaction time and movement time at 12 weeks
  Effect of 12 weeks treatment with iGlarLixi or Glargine on cognitive function assessed by established Reaction Time (RTI). Outcome measures: Reaction time and movement time for both the simple and five-choice variants.
  It is part of Cambridge Neuropsychological Test Automated Battery (CANTAB) to assess neurocognition. All CANTAB tests are evaluated together.
Cognitive function | Change from baseline latency, probability of false alarms and sensitivity at 12 weeks
  Effect of 12 weeks treatment with iGlarLixi or Glargine on cognitive function assessed by established Rapid Visual Information Processing (RVP). Outcome measures: Latency (speed of response), probability of false alarms and sensitivity.
  It is part of Cambridge Neuropsychological Test Automated Battery (CANTAB) to assess neurocognition. All CANTAB tests are evaluated together.
Cognitive function | Change from errors made by the participant, the number of trials required to locate the pattern(s) correctly, memory scores and stages completed baseline at 12 weeks
  Effect of 12 weeks treatment with iGlarLixi or Glargine on cognitive function assessed by established Paired Associates Learning (PAL). Outcome measures: Errors made by the participant, the number of trials required to locate the pattern(s) correctly, memory scores and stages completed.
  It is part of Cambridge Neuropsychological Test Automated Battery (CANTAB) to assess neurocognition. All CANTAB tests are evaluated together.
Cognitive function | Change from baseline errors and strategy at 12 weeks
  Effect of 12 weeks treatment with iGlarLixi or Glargine on cognitive function assessed by established Spatial Working Memory (SWM). Outcome measures: errors (selecting boxes that have already been found to be empty and revisiting boxes which have already been found to contain a token) and strategy.
  It is part of Cambridge Neuropsychological Test Automated Battery (CANTAB) to assess neurocognition. All CANTAB tests are evaluated together.
Cognitive function | Change from baseline number and percentage of correct trials and latency at 12 weeks
  Effect of 12 weeks treatment with iGlarLixi or Glargine on cognitive function assessed by established Pattern Recognition Memory (PRM). Outcome measures: Number and percentage of correct trials and latency (speed of participant's response) It is part of Cambridge Neuropsychological Test Automated Battery (CANTAB) to assess neurocognition. All CANTAB tests are evaluated together.
Cognitive function | Change from baseline latency, the number of correct patterns selected and a statistical measure giving the probability of an error after a correct or incorrect response at 12 weeks
  Effect of 12 weeks treatment with iGlarLixi or Glargine on cognitive function assessed by established Delayed Matching to Sample (DMS). Outcome measures: Latency (the participant's speed of response), the number of correct patterns selected and a statistical measure giving the probability of an error after a correct or incorrect response.
  It is part of Cambridge Neuropsychological Test Automated Battery (CANTAB) to assess neurocognition. All CANTAB tests are evaluated together.
Glycemic control | Change from baseline glycemic control at 12 weeks
  Effect of 12 weeks treatment with iGlarLixi or Glargine on glycemic control (HbA1c change from baseline to week 12.
Liver fat content | Change from baseline body fat distribution at 12 weeks
  Will be assessed by liver MR-spectroscopy change from baseline to 12 weeks.Unit: [%]
Total adipose tissue (TAT) | Change from baseline body fat distribution at 12 weeks
  Will be assessed by whole body MRI as change from baseline to 12 weeks. Unit: [l]
Visceral adipose tissue (VAT) | Change from baseline body fat distribution at 12 weeks
  Will be assessed by whole body MRI as change from baseline to 12 weeks. Unit: [l]
Subcutaneous adipose tissue (SCAT) | Change from baseline body fat distribution at 12 weeks
  Will be assessed by whole body MRI as change from baseline to 12 weeks. Unit: [l]
Body fat | Change from baseline body fat at 12 weeks
  Will be assessed by bioelectric impedance analysis (BIA) as change from baseline to 12 weeks. Unit: [%]
Lean body mass | Change from baseline body fat at 12 weeks
  Will be assessed by bioelectric impedance analysis (BIA) as change from baseline to 12 weeks. Unit: [kg]
Body weight | Change from baseline body weight at 12 weeks
  Will be assessed as change from baseline to 12 weeks. Unit [kg]

OTHER OUTCOMES:
Hypoglycemia | 1 week, 2 weeks, 4 weeks, 8 weeks and 12 weeks after randomisation
  Number of hypoglycemic events be recorded.
Hypoglycemia time of day | 1 week, 2 weeks, 4 weeks, 8 weeks and 12 weeks after randomisation
  Time of day for each hypoglycemic event (see therefore outcome 18) be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tuebingen, Department of Internal Medicine IV, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No